CLINICAL TRIAL: NCT07217405
Title: Low-Dose Radiotherapy Compared to Corticosteroid Injection for Treatment of Hand Osteoarthritis
Brief Title: Radiotherapy Compared to Corticosteroid Injection for Treatment of Hand Osteoarthritis
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Terin T. Sytsma, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24-010252
Record Dates: First submitted 2025-10-14; First posted 2025-10-16 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Osteoarthritis Hand; Osteoarthritis Wrist
MeSH Terms: interventions — Adrenal Cortex Hormones; Methylprednisolone; Lidocaine; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Low-dose radiotherapy (LDRT) (Experimental): Subjects will receive a total of six (6) low-dose radiotherapy (LDRT) treatments for hand osteoarthritis.
  Interventions: Radiation: Low-dose radiotherapy (LDRT)
- Corticosteroid injection (CSI) (Active Comparator): Subjects will receive standard of care corticosteroid injection (CSI) therapy for hand osteoarthritis.
  Interventions: Drug: Corticosteroid injection (CSI)

INTERVENTIONS:
Drug: Corticosteroid injection (CSI) — A maximum of 3 joints will be treated with standard a standard combination of methylprednisolone and lidocaine:
  * 1st Carpometacarpal (CMC) joint - 20 mg methylprednisolone/0.5 mL 1% lidocaine*
  * Radiocarpal (RC) joint - 40 mg methylprednisolone/1 mL 1% lidocaine*
  * Scaphotrapeziotrapezoidal (STT) joint - 20 mg methylprednisolone/0.5 mL 1% lidocaine*
  * Metacarpophalangeal (MCP) joint - 20 mg methylprednisolone/0.5 mL 1% lidocaine
  * Interphalangeal (IP) joint - 10 mg methylprednisolone/0.25 mL 1% lidocaine
  Other Names: Methylprednisolone; Lidocaine
  Arms: Corticosteroid injection (CSI)
Radiation: Low-dose radiotherapy (LDRT) — Subjects will be treated with low-dose radiotherapy of 300cGy in 6 fractions, 2-3 times per week on non-consecutive days.
  Non-responders to the initial LDRT treatment will receive a second treatment course of 300cGy in 6 fractions to be given 2-3 times per week on non-consecutive days.
  Arms: Low-dose radiotherapy (LDRT)

SUMMARY:
The purpose of this research is to compare low-dose radiotherapy to corticosteroid injection for treatment of hand/wrist osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* Patient at Mayo Clinic, Rochester, MN
* Age 50 years or older
* Mild, moderate, or severe hand OA (Kellgren and Lawrence classification grade 2, 3, or 4) on hand radiographs within the last 24 months
* Hand OA pain with a minimum VAS score relating to hand pain of ≥40 (on a 100-point scale) when using the affected hand
* Ability to complete study questionnaires

Exclusion Criteria:

* History of previous surgery to the affected hand(s)
* Autoimmune joint disease such as rheumatoid arthritis or psoriatic arthritis
* Active confounding hand condition such as stenosing tenosynovitis or Dupuytren's contracture
* Recent injury (within last 1 month) to the affected hand causing current pain
* History of crystalline arthritis (gout or pseudogout) flare in the affected hand(s)
* Active use of opioid pain medication(s) or oral steroids within the last 3 months
* Fibromyalgia or central sensitization syndrome
* Hand CSI or other hand injection within the past 3 months
* History of hand LDRT within the past 3 months
* Poorly controlled diabetes (HbA1c > 10%)
* Active infection
* Current pregnancy

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Estimated)
Dates: Start 2025-12-23 (Estimated); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Change in Visual Analog Scale (VAS) score | Baseline, monthly for 6 months post-intervention, 9 months post-intervention, 12 months post-intervention
  Pain values reported by participants will be assessed using the 100-mm Visual Analogue Scale (VAS). The VAS line will be 100 mm long with no intermediate delineations. Each end will be marked with "no pain" on the left, and "worst possible pain" on the right. Participants will identify their pain level by indicating a point on the line between each end. That point will be measured from the "No pain" end, and the number of millimeters will be reported as the pain score.

SECONDARY OUTCOMES:
Change in Cochin Hand Function Scale scores | Baseline, monthly for 6 months post-intervention, 9 months post-intervention, 12 months post-intervention
  The Cochin Hand Function Scale (CHFS) uses an 18-item, 5-point Likert scale (0 to 5) for scoring, where higher scores indicate greater difficulty with hand function. Scores range from 0 (no difficulty) to 90 (impossible to complete) by summing the ratings for all 18 items. This scale measures the ability to perform daily activities related to the hand, such as kitchen tasks, dressing, and hygiene.
Change in analgesic medication use | Baseline, monthly for 6 months post-intervention, 9 months post-intervention, 12 months post-intervention
  Change in analgesic medication use will be assessed using the Qualitative Analgesic Questionnaire [QAC]. The QAC is a 3 question self-report survey tracking current use of pain medications.
Patient experience, as measured by Was It Worth It questionnaire | 6 months and 12 months post-intervention
  The Was It Worth It questionnaire is a 4-question survey consisting of yes/no questions regarding the treatment experience. The greater number of questions with a 'yes' response indicate a higher level of patient satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Terin Sytsma, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials